CLINICAL TRIAL: NCT02211924
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses (50 mg to 800 mg) of BI 44847 as Tablet(s) Administered to Healthy Male Subjects. A Randomised, Placebo-controlled (Within Dose Groups) and Double-blinded Trial
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BI 44847 Administered to Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1224.11
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (2):
- BI 44847 (Experimental): single rising dose
  Interventions: Drug: BI 44847
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 44847
  Arms: BI 44847
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to investigate safety, tolerability, pharmacokinetics and pharmacodynamics of BI 44847 in Japanese healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be healthy male volunteers who meet the criteria below:

  * Persons without clinically remarkable findings or clinically evident complications based on their concurrent illness, past medical history, physical examination, vital signs (blood pressure, pulse rate, and body temperature), 12-lead ECG, and laboratory test results
  * Persons who are 20 or older and 35 or younger
  * Persons with a BMI 18.5 kg/m2 or more and 25.0 kg/m2 less
  * Persons who are willing to participate in this trial before study initiation and who give their written consent in accordance with Good Clinical Practice

Exclusion Criteria:

* Any finding of the medical examination (including BP, Pulse Rate (PR) and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of any drugs within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within four months prior to administration or during the trial
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL) within four weeks prior to administration or during the trial
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre 19. A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome)
* The use of concomitant medications that prolong the QT/QTc interval
* Any ECG value outside of the reference range and of clinical relevance including, but not limited to QRS interval >120 ms
* Elevated urinary glucose levels at screening (>15 mg/dl)

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-08; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically relevant changes in vital signs | up to day 7
Number of patients with clinically relevant finding in 12-lead electrocardiogram (ECG) | up to day 7
Number of patients with clinically relevant changes in laboratory parameters | up to day 7
Number of patients with adverse events | up to 5 weeks

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | up to 48 hours after drug administration
tmax (time from dosing to maximum concentration) | up to 48 hours after drug administration
AUC0-inf. (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 48 hours after drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | up to 48 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 48 hours after drug administration
λz (terminal rate constant in plasma) | up to 48 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma | up to 48 hours after drug administration
MRTpo (mean residence time of the analyte in the body after po administration) | up to 48 hours after drug administration
CL/F (total clearance of the analyte in the plasma after extravascular administration) | up to 48 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 48 hours after drug administration
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2) | up to 48 hours after drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 48 hours after drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 48 hours after drug administration
Area under the plasma glucose concentration time curve | up to 12 hours after drug administration
Total amount of glucose excreted in the urine | up to 48 hours after drug administration
Maximum glucose concentration in plasma | up to 12 hours after drug administration
Maximum glucose concentration in urine | up to 48 hours after drug administration